CLINICAL TRIAL: NCT06071988
Title: Long Term Efficacy and Tolerability of AP707 in Patients With Chronic Pain Due to Traumatic or Post-operative Peripheral Neuropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Apurano Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DISCOVER__(PNP2)
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-09

CONDITIONS: Pain; Pain Syndrome; Pain, Chronic; Chronic Pain; Chronic Pain Syndrome; Neuropathic Pain; Peripheral Neuropathy; Peripheral Neuralgia; Peripheral Nerve Injury; Post Operative Pain; Post-Traumatic Neuralgia; Plexopathy
Keywords: Adezunap; Pain Therapy; Pain; Pain Syndrome; Chronic Pain; Chronic Pain Syndrome; Peripheral Nervous System; PNS; Neuropathic Pain; Peripheral Neuropathy; Peripheral Neuralgia; Peripheral Nerve Injury; Post Operative Pain; Post-Traumatic Neuralgia; Plexopathy; THC; Tetrahydrocannabinol; Delta-9-Tetrahydrocannabinol; Cannabis; Cannabinoids
MeSH Terms: conditions — Pain; Somatoform Disorders; Chronic Pain; Neuralgia; Peripheral Nervous System Diseases; Peripheral Nerve Injuries; Pain, Postoperative; Agnosia; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Sublingual spray with maximum application of 16 actuations per day or a maximum daily dose of 17,6mg THC distributed over 4 daily intakes.
  Interventions: Drug: Adezunap (AP707)
- Control group (Experimental): Sublingual spray with maximum application of 16 actuations per day distributed over 4 daily intakes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adezunap (AP707) — Sublingual spray with maximum application of 16 actuations per day or a maximum daily dose of 17,6mg THC distributed over 4 daily intakes.
  Arms: Treatment group
Drug: Placebo — Sublingual spray with maximum application of 16 actuations per day distributed over 4 daily intakes.
  Arms: Control group

SUMMARY:
Over the last years a rising medical need for treatment of chronic pain was identified. Based on previous findings indicating the pain modulating effects of cannabinoids in chronic pain disorders, this clinical trial investigates the long term efficacy and tolerability of the THC-focused nano endocannabinoid system modulator AP707 in patients with chronic pain disorders due to traumatic or post-operative peripheral neuropathy. Patients receive AP707 or placebo over the course of 14 weeks as an add-on to the standard of care. Changes in pain intensity, quality of life and sleep and others measures are monitored through different scales to assess the efficacy of AP707 in patients with chronic pain due to traumatic or post-operative peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Patients with chronic pain due to traumatic or post-operative peripheral neuropathy since at least 3 months
3. Female and male patients (> 18 years)
4. Patients with more than 1 year life expectancy
5. Patients with optimized sCPT on study entry as defined in section 3.1.1 and section 3.1.3 of the study protocol
6. Willingness of study patients of both sexes to use reliable contraception during study participation and for three months after taking the last study medication
7. Good command of German language, in order to understand questionnaires in German
8. Current moderate to severe pain with pain intensity > 5 on Numeric Rating Scale (NRS, 0 - 10) and thus an existing need for further pain therapy
9. Completed QUISS (Quantification Inventory for Somatoform Syndromes) questionnaire with 45 or less score points

Exclusion Criteria:

1. Medical history of hypersensitivity or intolerance to the investigational product or its ingredients or to ingredients of similar chemical structure
2. Known intolerance to cannabinoids or cannabis products.
3. Participation in another clinical trial within the last four weeks prior to inclusion.
4. Pregnant or nursing women (as excluded by pregnancy testing at visit 1).
5. Other medical conditions that do not allow the trial subject to appraise the nature, scope, and potential consequences of the clinical trial
6. Indications that the trial subject is unlikely to comply with the study protocol (e.g., unwillingness to cooperate)
7. Known use of medicinal cannabis products within the last 8 weeks
8. Active malignant tumor disease, tumor pain, or other dominant severe pain other than that of the study indication
9. Known history of severe liver or kidney diseases
10. Known history of severe cardiovascular disease
11. Known history of or acute mental illness such as severe depression, psychosis, bipolar disorder, mania, anxiety, or obsessive-compulsive disorder
12. Known history of addictive disease (e.g., alcohol, medication, drug addiction)
13. Answered during Screening less than 12 times of 18 the pain intensity (NRS) inquiry
14. Laboratory liver values: Alanine aminotransferase (ALT, GPT) > 3 x ULN (Upper Limit of Normal range), Aspartate aminotransferase (AST, GOT) > 3 x ULN, Alkaline phosphatase (AP) > 2.5 x ULN, and for bilirubin > 1.5 x ULN
15. Laboratory renal value: Serum creatinine > 1.5 ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain level on the Numeric Rating Scale (NRS, 0-10) between baseline and at treatment week 14 (end of first treatment phase) in comparison of study arm 1 (verum) and study arm 2 (placebo) | Once daily in week 4 and 14

SECONDARY OUTCOMES:
Change in pain level on the Numeric Rating Scale (NRS, 0-10) between baseline and at treatment week 26 (end of second treatment phase) in comparison of study arm 1 (verum) and study arm 2 (placebo) | Once daily in week 4 and 26
Change in pain level on the Numeric Rating Scale (NRS, 0-10) between baseline and at treatment week 52 (end of third treatment phase) in comparison of study arm 1 (verum) and study arm 2 (placebo) | Once daily in week 4 and 52
Change in the pain score of the Neuropathic Pain Symptom Inventory (NPSI) questionnaire between baseline and at treatment week 14, treatment week 26 and treatment week 52 in comparison of study arm 1 (verum) and study arm 2 (placebo) | Once in week 1, 14, 26 and 52
Change in pain level on the Numeric Rating Scale (0-10) between baseline and in treatment week 5, 11, 18, 22, 30, 34, 43, 47 in comparison of study arm 1 (verum) and study arm 2 (placebo) | Several times weekly in week 4, 5, 11, 18, 22, 30, 34, 43 and 47
Responder analysis for endpoints 1), 2), 3) and 4) for treatment week 14, 26 and 52 | Week 14, 26 and 52
  1. Proportion of patients who experienced > 30 % improvement in pain score (Numeric Rating Scale)
  2. Proportion of patients who experienced > 40 % improvement in pain score (Numeric Rating Scale)
  3. Proportion of patients who experienced > 50 % improvement in pain score (Numeric Rating Scale)
Change in sCPT (percentage of change in dosage and percentage of change in combination of analgesic measures) in both study arms from start to week 14 | Week 14
Change in psychological distress using Depression Anxiety Stress Scales Short Form (DASS-21) questionnaire from start to week 14, 26, and 52 | Week 1, 14, 26 and 52
Change of Patient Global Impression of Change (PGIC) from start to week 14, 26, and 52 | Week 14, 26 and 52
Change in quality of life using the Veterans RAND (VR-12) questionnaire from start to week 14, 26, and 52 | Week 1, 14, 26 and 52
Change in sleep quality using the Regensburg Insomnia Scale (RIS) from start to week 14, 26, and 52 | Week 1, 14, 26 and 52
Change in pain score of the Brief Pain Inventory - Short Form (BPI-SF) questionnaire from start to week 14, 26, and 52 | Week 1, 14, 26 and 52
Area under NRS-curve until treatment week 5, 11, 14, 18, 22, 26, 30, 34, 39, 43, 47, 52 | Week 5, 12, 18, 22, 26, 30, 34, 39, 43, 47 and 52
Change in VR-12 components (physical component summary PCS, mental component summary MCS) from start to week 14, 26, and 52 | Week 1, 14, 26 and 52
Number of patients with rescue medication over the course of the clinical trial and within periods: until treatment week ≤5, ≤11, ≤14, ≤18, ≤22, ≤26, ≤30, ≤34, ≤43, ≤47, ≤52 | Week 5, 11, 14, 18, 22, 26, 30, 34, 43, 47 and 52

OTHER OUTCOMES:
Number and severity of adverse events (AE) | Week 1 to 52

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Rechts der Isar (Zentrum für Interdisziplinäre Schmerztherapie), Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No